CLINICAL TRIAL: NCT00077753
Title: A Double-Blind, Placebo-Controlled, Parallel, Multicenter Study on Extended VTE Prophylaxis in Acutely Ill Medical Patients With Prolonged Immobilization
Brief Title: EXCLAIM:Extended Prophylaxis for Venous ThromboEmbolism (VTE) in Acutely Ill Medical Patients With Prolonged Immobilization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XRP4563C_3501
Record Dates: First submitted 2004-02-12; First posted 2004-02-16 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — enoxaparin sodium

INTERVENTIONS:
Drug: enoxaparin sodium

SUMMARY:
Primary objective:

* To demonstrate the superiority of extended VTE prophylaxis with enoxaparin 40mg sc qd for 28 ± 4 days, compared to placebo, both following 10 ± 4 days of initial treatment with enoxaparin 40mg sc qd

Secondary objectives:

* To assess the reduction in mortality rate at the end of the double-blind treatment period, at 3 (90 ± 10 days) and at 6 (180 ± 10 days) months from the time of entry to the study, in patients on extended prophylaxis
* To assess the incidence of VTE at 3 months (90 ± 10 days) from the time of randomization to the study
* To evaluate the safety of extended enoxaparin VTE prophylaxis in acutely ill medical patients with prolonged immobilization. Safety evaluation includes:

  * Major and minor hemorrhage
  * Heparin induced thrombocytopenia
  * Serious adverse events
* To assess differences in levels of health-care utilization and cost between patients receiving extended VTE prophylaxis versus those receiving placebo.

ELIGIBILITY:
Inclusion criteria:

* Recent immobilization ≤ 3 days
* Level 1 mobility patients who are ≥ 40 years of age with acute medical illness or acute exacerbation of chronic medical illness
* Level 2 mobility patients who

  * are >75 yrs of age
  * are ≥ 40 years of age and have a history of VTE (deep venous thrombosis or pulmonary embolism)
  * are ≥ 40 years of age and have a baseline diagnosis of cancer (active cancer or history of cancer)

Anticipated decreased level of mobility of 5 ± 2 days with a level of activity 1 and 2 at the time of study entry and likely to continue at a lower than pre-morbid activity level after the initial 5 ± 2 day period. PATIENTS DO NOT HAVE TO BE HOSPITALIZED IN ORDER TO BE INCLUDED IN THE STUDY.(Definition of decreased level of mobility: _Level 1:bed rest or sedentary patients _Level 2:level 1 with bathroom privileges)

* Presence of at least one of the following medical conditions:

  * Heart Failure, NYHA class III and IV

    * Class III : Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitationdyspnea, or anginal pain.
    * Class IV : Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
  * Acute respiratory insufficiency
  * Other acute medical conditions such as:

    * Acute ischemic stroke, any territory, with an appropriate neuroradiologic (head CT scan or brain MRI scan) providing results consistent with non hemorrhagic stroke
    * acute infection without septic shock
    * acute rheumatic disorders
    * active episode of inflammatory bowel disease
    * active cancer defined as history of histologically or cytologically confirmed cancer in patients who are not candidates for debulking or curative intent surgery at study entry
    * Any other acute medical illness or exacerbation of chronic medical illness resulting in clinically significant reduction in mobility as compared to premorbid level.

Exclusion criteria:

* Women who are breastfeeding, pregnant or of childbearing age and not using medically acceptable effective contraception
* Patients with any evidence of an active bleeding disorder
* Contraindication to anticoagulation
* Major surgery within the previous 3 months
* Patients who have had spinal or epidural analgesia or lumbar puncture within the preceding 24 hours
* Known hypersensitivity to heparin, or LMWH, or pork derived products
* A documented previous episode of heparin-induced or LMWH induced thrombocytopenia and/or thrombosis (HIT, HAT, or HITTS)
* Patients who have taken part in another clinical trial within the previous thirty days
* Patients with a persistent renal failure. The patient's creatinine level must be less than the creatinine level per gender/age/weight. This will replace the calculated creatinine clearance
* Known or suspected severe anemia of unexplained cause considered clinically relevant by investigator
* Patients with prosthetic heart valves
* Patients with known cerebral metastases

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4726
Dates: Start 2002-02; Primary Completion 2006-10 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
During double blind treatment : Cumulative occurrence of VTE assessed by ultrasound for all patients at 28±4 days after randomization (or earlier if symptomatic VTE) and/or V/Q lung scan for symptomatic patients ; Major hemorrhagic complications.

SECONDARY OUTCOMES:
Occurrence of VTE between Day 1 and Day 90±10, Mortality at the end of Double-Blind Treatment, at 3 and 6 months
Minor plus major hemorrhagic complications during Double-Blind Treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Sagnard, Study Director — Sanofi
Locations (20):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Buenos Aires, Argentina
- Sanofi-Aventis, North Ryde, Australia
- Sanofi-Aventis, Vienna, Austria
- Sanofi-Aventis, Brussels, Belgium
- Sanofi-Aventis, São Paulo, Brazil
- Sanofi-Aventis, Laval, Canada
- Sanofi-Aventis, Bogotá, Colombia
- Sanofi-Aventis, Paris, France
- Sanofi-Aventis, Berlin, Germany
- Sanofi-Aventis, Mumbai, India
- Sanofi-Aventis, Netanya, Israel
- Sanofi-Aventis, Milan, Italy
- Sanofi-Aventis, México, Mexico
- Sanofi-Aventis, Warsaw, Poland
- Sanofi-Aventis, Moscow, Russia
- Sanofi-Aventis, Johannesburg, South Africa
- Sanofi-Aventis, Barcelona, Spain
- Sanofi-Aventis, Mégrine, Tunisia
- Sanofi-Aventis, Guildford, United Kingdom

REFERENCES:
- [Derived] Chi G, Goldhaber SZ, Kittelson JM, Turpie AGG, Hernandez AF, Hull RD, Gold A, Curnutte JT, Cohen AT, Harrington RA, Gibson CM. Effect of extended-duration thromboprophylaxis on venous thromboembolism and major bleeding among acutely ill hospitalized medical patients: a bivariate analysis. J Thromb Haemost. 2017 Oct;15(10):1913-1922. doi: 10.1111/jth.13783. Epub 2017 Sep 4. PMID 28762617
- [Derived] Turpie AG, Hull RD, Schellong SM, Tapson VF, Monreal M, Samama MM, Chen M, Yusen RD; EXCLAIM Investigators. Venous thromboembolism risk in ischemic stroke patients receiving extended-duration enoxaparin prophylaxis: results from the EXCLAIM study. Stroke. 2013 Jan;44(1):249-51. doi: 10.1161/STROKEAHA.112.659797. Epub 2012 Nov 1. PMID 23117723
- [Derived] Sharma A, Chatterjee S, Lichstein E, Mukherjee D. Extended thromboprophylaxis for medically ill patients with decreased mobility: does it improve outcomes? J Thromb Haemost. 2012 Oct;10(10):2053-60. doi: 10.1111/j.1538-7836.2012.04874.x. PMID 22863355
- [Derived] Hull RD, Schellong SM, Tapson VF, Monreal M, Samama MM, Nicol P, Vicaut E, Turpie AG, Yusen RD; EXCLAIM (Extended Prophylaxis for Venous ThromboEmbolism in Acutely Ill Medical Patients With Prolonged Immobilization) study. Extended-duration venous thromboembolism prophylaxis in acutely ill medical patients with recently reduced mobility: a randomized trial. Ann Intern Med. 2010 Jul 6;153(1):8-18. doi: 10.7326/0003-4819-153-1-201007060-00004. PMID 20621900